CLINICAL TRIAL: NCT05037201
Title: A Randomized Trial of Text Message-Based Nudges to Increase COVID-19 Vaccination
Brief Title: Text Message Nudges for COVID-19 Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mitesh Patel (Industry)
Responsible Party: Sponsor-Investigator, Mitesh Patel, VP, Ascension, Ascension Health
Organization: Ascension Health (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RAS20210002
Record Dates: First submitted 2021-09-07; First posted 2021-09-08 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): The control arm will receive usual health system messaging about the importance and deadlines for receiving COVID-19 vaccination.
- Text message (Experimental): The intervention arm will receive a text message stating that the vaccine is reserved for them on a specific date. They will have the ability to reschedule to a different day, opt-out of this text messaging intervention, or if previously vaccinated they can upload documentation to the Ascension website.
  Interventions: Behavioral: Text message

INTERVENTIONS:
Behavioral: Text message — The intervention arm will receive a text message stating that the vaccine is reserved for them on a specific date. They will have the ability to reschedule to a different day, opt-out of this text messaging intervention, or if previously vaccinated they can upload documentation to the Ascension website.
  Arms: Text message

SUMMARY:
The COVID-19 pandemic has caused significant morbidity and mortality across the world. Effective vaccines are now available but underutilized. In July 2021, Ascension Health implemented a mandate requiring all employees to obtain the COVID-19 vaccine by November 12th. In August 2021, the number of COVID-19 cases in the US increased rapidly, specifically in states with lower vaccination rates, many of which are served by Ascension Health facilities. In this study, we will evaluate a rapidly deployed health system initiative to use text messaging to nudge Ascension employees who have not yet been vaccinated to commit to a date and receive vaccination.

DETAILED DESCRIPTION:
The COVID-19 pandemic has caused significant morbidity and mortality across the world. Effective vaccines are now available but underutilized. In July 2021, Ascension Health implemented a mandate requiring all employees to obtain the COVID-19 vaccine by November 12th. In August 2021, the number of COVID-19 cases in the US increased rapidly, specifically in states with lower vaccination rates, many of which are served by Ascension Health facilities.

Nudges are subtle changes to the way information is framed or choices are offered that can have a significant impact on behavior. Status quo bias is a preference for the current state which is often used as a reference point when making decisions. Changes from the reference point are often faced with high inertia and this prevents changes in behavior. Default options are the setting of the baseline reference point and are often taken as an implicit recommendation. In prior work, changing default options has led to significant changes in health-related behaviors. For example, changing prescription default settings in the EHR from opt-in to opt-out for generic prescriptions increased the rate of generic prescriptions from 75% to 98% across Penn Medicine (Patel et al. Annals of IM. 2014; Patel et al. JGIM 2018). Framing program participation as opt-out has led to a 22% increase in enrollment in a COVID-19 surveillance testing program (Oakes et al. NEJM Catalyst 2021) and triple enrollment in remote monitoring programs for medication adherence (Mehta et al. JAMA Cardiology. 2018) and diabetes management (Aysola et al. AJHP 2016)

ELIGIBILITY:
Inclusion Criteria:

* Ascension Associate Employee

Exclusion Criteria:

* Prior vaccination for COVID-19
* Exemption from COVID-19 vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Percent receiving COVID-19 Vaccine | 2 weeks
  The percent of participants that receive the COVID-19 vaccine within 2 weeks of the intervention.

SECONDARY OUTCOMES:
Time to receive COVID-19 vaccine | 4 weeks
  Time to COVID-19 vaccination in days within 4 weeks of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, Principal Investigator — Ascension
Locations (1):
- Ascension, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared

REFERENCES:
- [Derived] Patel MS, Fogel R, Winegar AL, Horseman C, Ottenbacher A, Habash S, Dukes JL, Brinson TC, Price SC, Masoudi FA, Cacchione J, Yehia BR. Effect of Text Message Reminders and Vaccine Reservations on Adherence to a Health System COVID-19 Vaccination Policy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2222116. doi: 10.1001/jamanetworkopen.2022.22116. PMID 35857327